CLINICAL TRIAL: NCT06688838
Title: Exploring the Clinical Features and Factors Related to Efficacy in Blau Syndrome: A Retrospective Observational Study
Brief Title: Effective Treatment of Jak1/3 Inhibitor in Blau Syndrome
Acronym: inapplicable
Status: Enrolling by invitation | Type: Observational
Sponsor: Tongji Hospital (Other)
Collaborators: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); Affiliated Hospital of Yunnan University (Other); Pfizer (Industry); Wuhan Women and Children's Medical Center (Other); Johns Hopkins Community Physicians (Other)
Responsible Party: Principal Investigator, YIKAI YU, associate chief physician, Tongji Hospital
Other Study IDs: TJ-IRB202409051; 201271031432 (Other Grant/Funding Number: Wuhan Scientific Funding for young investigators)
Record Dates: First submitted 2024-11-10; First posted 2024-11-14 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Blau Syndrome
Keywords: Blau syndrome; retrospective; Janus kinase inhibitors
MeSH Terms: conditions — Blau syndrome | interventions — tofacitinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (3):
- glucocorticoid+ DMARDs: glucocorticoid+ DMARDs
- glucocorticoid+TNFi: glucocorticoid+TNFi
- glucocorticoid+Tofacitinib: glucocorticoid+Tofacitinib
  Interventions: Drug: Tofacitinib

INTERVENTIONS:
Drug: Tofacitinib — If a patient does not respond well to DMARDs treatment, then Tofacitinib or TNFi treatment may be used instead.
  Other Names: TNFi
  Groups: glucocorticoid+Tofacitinib

SUMMARY:
To investigate the effectiveness of the JAK 1/3 inhibitor tofacitinib in treating Blau syndrome and explore the association between various clinical and genetic features and therapeutic responses within the cohort.

DETAILED DESCRIPTION:
Blau Syndrome (BS) is a monogenic systemic autoinflammatory disease characterized by dominantly inherited granulomatous inflammation due to mutations in nucleotide-binding oligomerization domain 2 gene (NOD2). Traditionally associated with a clinical trial of arthritis, dermatitis, and uveitis, recent observations have expanded its recognized manifestations to include systemic inflammatory features, skin or cutaneous vasculitis, and multi-organ involvement. Despite the rarity of BS, significant advances have been made through multi-center collaborations. Current studies, primarily retrospective, highlight the clinical diversity of BS, including cases with disease-causing NOD2 mutations but lacking the typical clinical trial . In response to gaps in understanding of BS's pathogenic mechanisms, the investigators initiated a retrospective observational study to collect detailed clinical data and perform whole exome sequencing, specifically targeting NOD2 mutations and STAT3 rs2293152 phenotypic variations to explore their relationships with therapeutic responses.

ELIGIBILITY:
Inclusion Criteria:

1. The patient must conform to the characteristic triad of granulomatous arthritis, uveitis, and dermatitis, or the characteristic non-caseous granuloma of BS indicated by skin or synovial biopsy;
2. Whole exon detection indicated characteristic mutations of NOD2 gene

Exclusion Criteria:

1. Patients with autoimmune diseases, including but not limited to lupus erythematosus, Sjogren's syndrome, vasculitis, ankylosing spondylitis, myositis, dermatomyositis, rheumatoid arthritis, etc.;
2. combined with other neoplastic diseases, such as lymphoma, leukemia, etc.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Retrieve patients diagnosed with Blau syndrome from the medical record system between January 2017 and December 2023.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
clinical responses | through study completion, an average of 1 year
  Inefficacy,Partial response, Good response,Clinical remission

CONTACTS AND LOCATIONS:
Locations (1):
- Yikai YU, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No
Not shared. Contact the researcher if necessary.

REFERENCES:
- [Derived] Hu Y, Li P, Liu J, Zeng Z, Zhang X, Yin W, Xu H, Cai J, Yu Y. Effective Treatment of Janus Kinase 1/3 Inhibitor in Blau Syndrome From a Multicenter Retrospective Study in Central China. J Rheumatol. 2025 Aug 1;52(8):810-816. doi: 10.3899/jrheum.2024-0822. PMID 40233998